CLINICAL TRIAL: NCT06887244
Title: Evaluation of the Effectiveness of Nurse Tele-consultation on the Quality of Elective Colonoscopy, Procedure-related Anxiety, and Financial Toxicity
Brief Title: Effectiveness of Nurse Tele-consultation on the Quality of Elective Colonoscopy, Procedure-related Anxiety, and Financial Toxicity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Registry 26-23
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Patient Satisfaction and Efficacy of Bowel-preparation; Colon Cancer Prevention
Keywords: colonoscopy; tele-consultation procedure; colon cancer; financial toxicity; anxiety procedure-related
MeSH Terms: conditions — Patient Satisfaction; Colonic Neoplasms; Financial Stress

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nurse tele-consultation arm (Experimental): Use of the nurse tele-consultation tool in the Intervention arm administered 5±2 days before the colonoscopy procedure.
  Interventions: Other: Tele-consultation
- Standard arm (No Intervention)

INTERVENTIONS:
Other: Tele-consultation — Tele-consultation procedure is defined as a telephone consultation with the patient conducted by nursing staff with an appropriate level of experience in digestive endoscopy
  Arms: nurse tele-consultation arm

SUMMARY:
This is a multicenter, non-pharmacological, experimental, prospective, randomized study, with two arms (1:1) in a single-blind design. The study aims to evaluate the effectiveness of a tele-consultation procedure in patients undergoing elective colonoscopy in terms of quality of the exam, anxiety procedure-related and financial toxicity.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness, in daily clinical practice, of a tele-consultation procedure (defined as a telephone consultation with the patient conducted by nursing staff with an appropriate level of experience in digestive endoscopy) with the goal of:

1. improving adherence to methods and timing for the correct intake of the intestinal preparation by patients undergoing elective colonoscopy;
2. assessing whether the tele-consultation can reduce anxiety and procedure-related stress, promoting a better emotional state in patients undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for outpatient pancolonoscopy:

* for diagnostic purposes;
* for screening purposes;
* for post-polypectomy follow-up;
* of both genders;
* of all ethnicities;

Exclusion Criteria:

* Patients under 18 years of age or over 80 years of age;
* Patients on waiting lists with SHORT priority: the procedure to be provided within a short time (no more than 10 days);
* Patients included in GOM pathways who undergo colonoscopy within 10 days;
* Pregnancy;
* Presence of known contraindications to bowel preparation;
* Presence of known contraindications to performing pancolonoscopy;
* Patients who have undergone colonic resection and/or have a colostomy/ileostomy;
* Patients with cognitive impairments;
* Patients declared legally incompetent or unable to understand and make decisions;
* Patients unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of intestinal preparation. BBPS score (BOSTON BOWEL PREPARATION SCORE) | at the end of colonoscopy up to 12 months
  Compare the quality of the colonoscopy between patients who received tele-consultation (INTERVENTION Group) and those who did not receive tele-consultation (CONTROL Group) based on the BBPS score (BOSTON BOWEL PREPARATION SCORE). The BBPS score ranges from 0 to 9 based on intestinal preaparation in cecum, colon and rectum. Each section is scored on a scale of 0 to 3 (0= unprepared to 3= excellent). The total BBPS score is the sum of the scores from the three sections (score 0 to 5=Poor preparation; score 6 to 7= fair preparation; score 8 to 9=good preparation). A higher score indicates better bowel preparation, which is ideal for a successful colonoscopy.
H.A.D.S. (Hospital Anxiety and Depression Scale) | baseline, before colonoscopy up to 12 months
  Compare the quality of the emotional state between the sample of patients who received tele-consultation (INTERVENTION Group) and those who did not receive tele-consultation (CONTROL Group) based on the H.A.D.S. score (Hospital Anxiety and Depression Scale).The scale consists of 14 items, with 7 questions related to anxiety and 7 related to depression. Each item is rated on a 4-point scale (from 0=not at all to 3= most of the time). The total score for each section (anxiety and depression) can range from 0 to 21, and then the scores from both sections are combined for a total score ranging from 0 to 42.
  The minimun score is 0-7 that means normal (little to no anxiety or depression). The maximum score is 15-21 that means severe (significant anxiety or depression).

SECONDARY OUTCOMES:
Financial Toxicity (FT) using the "PROFFIT questionnaire" | baseline (before colonoscopy) up to 12 months
  Assessment of FT through PROFFIT questionnaire. This is an Italian instrument for evaluating FT in patients in the Italian healthcare context. It includes 16 total items, 7 measuring FT (defining the PROFFIT financial score) and 9 measuring possible determinants of FT. The score range from 0-100 (the higher value means precence of FT).
Effectiveness of a colonoscopy in detecting adenomas. Adenoma Detection Rate (ADR) | at the end of colonoscopy up to 12 months
  Quality of colonoscopies between patients who received tele-consultation and those who did not receive tele-consultation based on ADR. ADR represents the percentage of patients undergoing colonoscopy in which at least one adenoma is detected.
Rate of cecal intubation | at the end of colonoscopy up to 12 months
  Cecal intubation rate in patients of the 2 study groups

CONTACTS AND LOCATIONS:
Overall Officials: Francesco De Falco, Nursing degree, Principal Investigator — National Cancer Institute, IRCCS Fondazione G. Pascale
Locations (1):
- S.S.D. Garoenterologia ed Endoscopia Digestiva, Naples, Italy

IPD SHARING:
Plan to Share IPD: No